CLINICAL TRIAL: NCT00698126
Title: A Multicentre, Open Label, Nonrandomised, Non-interventional, Observational, Safety Study in Subjects Using Insulin Aspart (NovoRapid® ) or Soluble Human Insulin for the Treatment of Diabetes Mellitus the UPGRADE Study
Brief Title: Observational Study of Patients Using NovoRapid® or Soluble Human Insulin for Treatment of Type 2 Diabetes
Acronym: UPGRADE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-1897
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: soluble human insulin
- B
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: soluble human insulin — Observational study; use of the products as in the normal clinical practice conditions
  Other Names: Actrapid
  Groups: A
Drug: biphasic insulin aspart — Observational study; use of the products as in the normal clinical practice conditions
  Groups: B

SUMMARY:
This trial is conducted in Europe. The aim of this observational study is to evaluate the incidence of major hypoglycaemic episodes in patients with type 2 diabetes treated with NovoRapid® or Soluble Human Insulin under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Treatment with Insulin Aspart (NovoRapid®) or Soluble Human Insulin for minimum 3 months and maximum 3 years

Exclusion Criteria:

* Patients with an end-stage renal failure
* Patients with a serious liver disease
* Patients with concomitant malignant disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 2 diabetes who is already in treatment with insulin aspart or soluble human insulin will be included in the study
Sampling Method: Probability Sample
Enrollment: 4099 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Number of major hypoglycaemic events reported as serious adverse drug reactions | after 26 weeks

SECONDARY OUTCOMES:
Number of serious and non serious drug reactions | during 26 weeks
Number of serious adverse event | during 26 weeks
Number of all major (daytime and nocturnal) hypoglycaemic events | during 26 weeks
Number of major hypoglycaemic events related to omission of a meal after injection | during 26 weeks
Number of major hypoglycaemic events related to physical exercise of at least 30 min duration | during 26 weeks
Number of all minor (daytime and nocturnal) hypoglycaemic events during 4 weeks preceding each study visit | after 26 weeks
Weight and waist circumference change | during 26 weeks
Number of hypoglycaemia events in the two different treatment groups based on the HbA1c level | after 26 weeks
Quality of Life (QoL) | after 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Rome, Italy

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com